CLINICAL TRIAL: NCT07026903
Title: The Impact of CGM on Weight Reduction in Women With Overweight/Obesity Without Accompanying Chronic Diseases
Brief Title: The Impact of CGM on Weight Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Maja Cigrovski Berkovic, Associate Professor, MD, PhD, specialist in internal medicine, subspecialist in endocrinology and diabetes, University of Zagreb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 84
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Obesity and Overweight; the Study Will Focus on Weight Reduction Through Lifestyle Changes Aided by Insights From Continuous Glucose Monitoring
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: women living with overweight/obesity will be allocated to either a group with or without addition of continuous glucose monitoring (CGM) in addition to lifestyle intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- experimental-randomized to isCGM (Other): experimental arm- participants randomized to isCGM during the 3 months lifestyle intervention trial duration control arm-participants not randomized to isCGM during the 3 months lifestyle intervention trial duration
  Interventions: Behavioral: resistance exercise and calorie restrictive diet

INTERVENTIONS:
Behavioral: resistance exercise and calorie restrictive diet — experimental group will be randomized to isCGM during the lifestyle intervention trial while control group will participate in the same lifestyle intervention but will not use isCGM

SUMMARY:
The goal of this randomized control study is to learn if continuous glucose monitoring (CGM) can aid in weight loss in overweight/obese women with no other chronic condition. The primary hypothesis is that insights from CGM aid in greater weight loss, and the secondary hypothesis is that the use of CGM reduces the dropout rate from a three-month exercise program. Research will compare the results of weight loss after inclusion into 3 month physical exercise and diet counselling program between experimental group (women assigned to wear CGM) and control group (women without CGM). All participants will be included in the same physical exercise program with a fitness coach (3 times weekly for 60 minutes per sessions, three different resistance trainings), and will be given a calorie-controlled diet based on a weekly menu.

DETAILED DESCRIPTION:
In this prospective study lasting 3 months, a total of 40 participants are planned to be included. The sample size was calculated using the free G Power program. For differences within the group (before-after measurements, 2 measurements), the required number of participants in one group would be 16 (with a power of 0.8 and the calculated effect size based on previous research = 0.66). Considering that differences between two groups will also be observed, the calculation was made more conservatively, using a moderate effect size factor for ANOVA for repeated measures (within-between interaction), and with a minimum required power of 0.8 and an effect size of 0.25, the total number of required participants is 28, which means 14 per group, assuming three BMI measurements. Due to the potential dropout rate, the sample size was increased to 20 participants per group. Participants will be recruited upon enrollment at the fitness center. Participants will be randomly divided into two groups; one that will use isCGM (FreeStyle Libre 2) for glucose control and nutritional choices, and a group without CGM (the control group). At the beginning of the study, all participants will have their body composition measured on a scale, BMI, waist and hip circumference, triceps skinfold thickness, and blood samples taken for biochemical analyses (CBC, glucose, HbA1c, lipid profile, aminotransferases, fT4, and TSH). Blood tests will be analyzed in the private laboratory. Only those participants who do not have glucose metabolism disorders (prediabetes or diabetes), significant anemia, clinically manifest hypo- or hyperthyroidism, or recent musculoskeletal injuries that would limit their participation in the exercise program will be included in the further study. All participants will undergo nutritional counseling and receive a proposal for a calorie-controlled diet based on a weekly menu. Participants will be asked to keep a food diary. Additionally, all participants will follow the same exercise program for 3 months under the professional guidance of a kinesiologist. Exercise will be conducted 3 times a week for 60 minutes in groups of up to 5 participants, and will include three different training sessions with external and bodyweight resistance. In the case of external resistance, weights will be adjusted according to the participants' status so that they can complete the assigned number of repetitions, and in the case of bodyweight exercises, participants who cannot complete the prescribed series will be allowed to take breaks between repetitions. At the midpoint of the program, after 1.5 months of research, body composition will be re-evaluated on the scale, and measurements of the triceps skinfold and waist and hip circumference will be repeated. Participants assigned to the CGM group will wear sensors (FreeStyle Libre 2, Abbott) for 2 weeks three times during the study (at the beginning, after 1.5 months, and after 3 months). At the end of the program, anthropometric measurements and biochemical indicators will be repeated as at the beginning of the study. Data will only be analyzed for those participants who attend more than 90% of the exercise sessions. Dropout rates and participant satisfaction with the program will be monitored, knowledge of macronutrients will be compared before and after the program, and initial and control laboratory results and anthropometric measures will be compared.

ELIGIBILITY:
Inclusion Criteria: females, age over 18 years, overweight/obese

Exclusion Criteria: prediabetes/diabetes, significant anemia, clinically manifest hypo- or hyperthyroidism, recent musculoskeletal injuries that would limit participation in the exercise

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — females
Enrollment: 35 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
change from baseline in the body mass index and body composition | the study will last for 3 months
  we will measure, compare and report changes in body weight, BMI and body composition in women living with overweight/obesity allocated to lifestyle measures+CGM and lifestyle measures without CGM

SECONDARY OUTCOMES:
changes in drop out rate between women living with overweight/obesity allocated to lifestyle intervention+CGM and those on lifestyle intervention | the study will last for 3 months
  we hypothesize that addition of CGM to lifestyle intervention will improve the adherence rate

CONTACTS AND LOCATIONS:
Locations (1):
- Fitness centre "Fit by Ines", Čakovec, Croatia

IPD SHARING:
Plan to Share IPD: Undecided